CLINICAL TRIAL: NCT03462576
Title: Companion Protocol for the ¹³C-Methacetin Breath Test Using the BreathID® MCS System for Conatus Phase 2 Study of Emricasan, an Oral Caspase Inhibitor, Under Protocol IDN-6556-17
Brief Title: Companion Protocol for Methacetin Breath Test (MBT) in Conatus Protocol IDN-6556-17
Status: Terminated | Type: Interventional
Why Stopped: Sponsor of Trial decision
Sponsor: Meridian Bioscience, Inc. (Industry)
Collaborators: Conatus Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: CON-EX-0217
Record Dates: First submitted 2018-03-06; First posted 2018-03-12 (Actual); Results first posted 2020-12-16 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Decompensated Cirrhosis
MeSH Terms: interventions — 3-(2-(2-tert-butylphenylaminooxalyl)aminopropionylamino)-4-oxo-5-(2,3,5,6-tetrafluorophenoxy)pentanoic acid

STUDY DESIGN:
Intervention Model Description: The study treatment duration will be at least 48 weeks with study visits every 4 weeks up to Week 48 and every 8 weeks after Week 48. All subjects will continue treatment until the last subject in the study reaches 48 weeks in the study. At least 30% of subjects randomized should have baseline MELD score ≥15 and ≤20.
  For each subject, the study will consist of:
  * Screening period of up to 4 weeks
  * Randomized, double-blind treatment period of at least 48 weeks
  * A follow-up visit 2 weeks after completion of study drug treatment The duration of each subject's participation will be at least 54 weeks for those completing the entire study.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The collaborator is responsible for the masking process.
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (3):
- Emricasan 25mg (Experimental): The study treatment duration will be at least 48 weeks with study visits every 4 weeks up to Week 48 and every 8 weeks after Week 48.
  Interventions: Combination Product: Methacetin Breath Test; Drug: Emricasan
- Emricasan 5mg (Experimental): The study treatment duration will be at least 48 weeks with study visits every 4 weeks up to Week 48 and every 8 weeks after Week 48.
  Interventions: Combination Product: Methacetin Breath Test; Drug: Emricasan
- Placebo (Placebo Comparator): The study treatment duration will be at least 48 weeks with study visits every 4 weeks up to Week 48 and every 8 weeks after Week 48.
  Interventions: Combination Product: Methacetin Breath Test; Drug: Placebo oral capsule

INTERVENTIONS:
Combination Product: Methacetin Breath Test — A breath analyzer will be used to measure changes in carbon 12 to carbon13 ratio as a result of metabolism of the Methacetin substrate before and after treatment.
Drug: Emricasan — Investigational drug for NASH treatment in Main Conatus protocol
  Arms: Emricasan 25mg; Emricasan 5mg
Drug: Placebo oral capsule — Placebo versus emricasan in Conatus NASH treatment trial
  Arms: Placebo

SUMMARY:
This study is a companion protocol that will use the data generated by Conatus' study of emricasan under protocol IDN-6556-17.The IDN-6556-17 study is a Phase 2, multicenter, double-blind, placebo-controlled trial of Emricasan in subjects with decompensated non-alcoholic steatohepatitis (NASH) cirrhosis.

DETAILED DESCRIPTION:
The protocol is intended to validate the ability of the MBT to predict deterioration by 48 weeks for all subjects, and at later time points for those followed longer, for subjects with decompensated NASH cirrhosis in the placebo treatment arm of Conatus' study IDN-6556-17.

As one of the Conatus' study secondary objectives, this companion protocol is designed to assess improvement in liver metabolic function as measured by Methacetin Breath Test (MBT) [ Time Frame: Baseline - Final Treatment Visit (at least 48 weeks to a max of 120 weeks) ].

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 years or older, able to provide written informed consent and able to understand and willing to comply with the requirements of the study.
2. Cirrhosis due to NASH with exclusion of other causes of cirrhosis (e.g. chronic viral hepatitis, alcoholic liver disease, etc.)
3. At least one of the following: a) history of variceal hemorrhage (more than 3 months prior to day 1) documented on endoscopy and requiring blood transfusion, b) history of at least moderate ascites (on physical exam or imaging) currently treated with diuretics.
4. MELD score ≥12 and ≤20 during screening
5. Albumin ≥2.5 g/dL during screening
6. Serum creatinine ≤1.5 mg/dL during screening

Exclusion Criteria:

1. Evidence of severe decompensation
2. Non-cirrhotic portal hypertension
3. Child-Pugh score ≥10
4. Current use of anticoagulants that affect prothrombin time or international normalized ratio
5. ALT >3 times upper limit of normal (ULN) or AST >5 times ULN during screening
6. Initiation or discontinuation of non-selective beta blockers within 1 month of screening
7. Transjugular intrahepatic portosystemic shunt or other porto-systemic bypass procedure within 1 year of screening or previously requiring revision
8. Alpha-fetoprotein >50 ng/mL in the last year
9. History of hepatocellular carcinoma (HCC) or evidence of HCC
10. History of malignancies other than HCC, unless successfully treated with curative intent and believed to be cured
11. Prior liver transplant
12. Uncontrolled diabetes mellitus (HbA1c >9%)
13. Change in diabetes medications or vitamin E within 3 months of screening
14. Restrictive bariatric surgery or bariatric device within 1 year of screening or prior malabsorptive bariatric surgery
15. Symptoms of biliary colic unless resolved following cholecystectomy
16. History of significant alcohol consumption within the past 5 years
17. Current use of medications that are considered inhibitors of organic anion transporting polypeptide OATP1B1 and OATP1B3 transporters
18. Prolongation of screening (pre-treatment) QTcF interval of >500 msecs, or history or presence of clinically concerning cardiac arrhythmias
19. Significant systemic or major illness other than liver disease
20. Human immunodeficiency virus infection
21. Use of alcohol, controlled substances (including inhaled or injected drugs), or non-prescribed use of prescription drugs within 1 year of screening to the point of interfering with the subject's ability to comply with study procedures and study drug administration in the investigator's judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Florida Digestive Health Specialists Research Institute, Lakewood Rch, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 60 subjects were disqualified at baseline before being divided into arms due to screen failure.
Groups:
- Patients With Number of Subjects Experiencing a High Risk Event in 25 mg Treatment Arm: Arm 1. The number of subjects that experience a decompensation event as described in the protocol in the arm treated with 25 mg of Emricasan.
- Number of Subjects Experiencing a High Risk Event in 5 mg Treatment Arm: Arm 2. The number of subjects that experience a decompensation event as described in the protocol in the arm treated with 5 mg of Emricasan.
- Number of Subjects Experiencing a High Risk Event in Placebo Arm: Arm 3. The number of subjects that experience a decompensation event as described in the protocol in the placebo arm .
Period: Overall Study
Arm/Group | Patients With Number of Subjects Experiencing a High Risk Event in 25 mg Treatment Arm | Number of Subjects Experiencing a High Risk Event in 5 mg Treatment Arm | Number of Subjects Experiencing a High Risk Event in Placebo Arm
Started | 46 | 48 | 45
Completed | 41 | 37 | 37
Not Completed | 5 | 11 | 8
Not completed — Protocol Violation | 5 | 11 | 7
Not completed — Device Malfunction | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Number of Subjects Experiencing a High Risk Event in 25 mg Treatment Arm: Arm 1. The number of subjects that experience a decompensation event as described in the protocol in the arm treated with 25 mg of Emricasan.
- Total: Total of all reporting groups
Arm/Group | Number of Subjects Experiencing a High Risk Event in 25 mg Treatment Arm | Number of Subjects Experiencing a High Risk Event in 5 mg Treatment Arm | Number of Subjects Experiencing a High Risk Event in Placebo Arm | Total
Number analyzed (Participants) | 46 | 48 | 45 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 1 subject's test was discontinued due to device malfunction.
  years
    number analyzed (Participants) | 46 | 48 | 44 | 138
    (all) | 59.674 (9.307) | 60.875 (8.668) | 62.864 (7.135) | 61.1 (8.48)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 subject test was discontinued due to device malfunction.
  Participants
    number analyzed (Participants) | 46 | 48 | 44 | 138
    Female | 26 | 19 | 27 | 72
    Male | 20 | 29 | 17 | 66
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 1 subject test was discontinued due to device malfunction.
  Participants
    number analyzed (Participants) | 46 | 48 | 44 | 138
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 1 | 1 | 1 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 0 | 2 | 1 | 3
    White | 43 | 43 | 41 | 127
    More than one race | 1 | 2 | 1 | 4
    Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants] — Population: 1 subject test was discontinued due to device malfunction.
  Participants
    United States: number analyzed (Participants) | 46 | 48 | 44 | 138
    United States | 46 | 48 | 44 | 138

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Experiencing a High Risk Event Based on a 5.5%/Hour Cut-off
Description: Binary diagnosis of subjects that are at high risk to develop a deterioration event as determined by the Methacetin Breath Test (MBT) derived from an algorithm developed under other Exalenz clinical studies using a pre-designed cutoff of Percentage Dose Recovery (PDR) peak of < 5.5%/hour. The data was collected and analyzed agnostic to the intervention.
Time Frame: 1 hour for MBT for assessment of this diagnostic outcome assessed during screening
Population: The population analyzed is Intent to Diagnose (ITD)
Measure: Count of Participants; unit: Participants
Groups:
- Number of Subjects Experiencing a High Risk Event in Placebo Arm: Arm 3. The number of subjects that experience a decompensation event as described in the protocol in the placebo arm.
Arm/Group | Number of Subjects Experiencing a High Risk Event in 25 mg Treatment Arm | Number of Subjects Experiencing a High Risk Event in 5 mg Treatment Arm | Number of Subjects Experiencing a High Risk Event in Placebo Arm
Number analyzed (Participants) | 46 | 48 | 44
Participants
  Events in subjects below cut-off | 3 | 4 | 6
  No event recorded in subjects below cut-off | 1 | 2 | 5
  Events in subjects above cut-off | 15 | 14 | 11
  No event recorded in subjects above cut-off | 27 | 28 | 22

2. Secondary Outcome: Number of Subjects Experiencing a High Risk Event Based on a 7.5 %/Hour Cut-off
Description: Binary diagnosis of subjects that are at high risk to develop a deterioration event as determined by the Methacetin Breath Test (MBT) derived from an algorithm developed under other Exalenz clinical studies using a pre-designed cutoff of Percentage Dose Recovery (PDR) peak of < 7.5%/hour.The data was collected and analyzed agnostic to the intervention.
Time Frame: 1 hour for MBT for assessment of this diagnostic outcome assessed during screening
Population: The population analyzed is Intent to Diagnose (ITD).
Measure: Count of Participants; unit: Participants
Arm/Group | Number of Subjects Experiencing a High Risk Event in 25 mg Treatment Arm | Number of Subjects Experiencing a High Risk Event in 5 mg Treatment Arm | Number of Subjects Experiencing a High Risk Event in Placebo Arm
Number analyzed (Participants) | 46 | 48 | 44
Participants
  Events in subjects below cut-off | 4 | 8 | 9
  No event recorded in subjects below cut-off | 4 | 4 | 6
  Events in subjects above cut-off | 14 | 10 | 8
  No event recorded in subjects above cut-off | 24 | 26 | 21

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for a period of 48 weeks
Arm/Group | Number of Subjects Experiencing a High Risk Event in 25 mg Treatment Arm | Number of Subjects Experiencing a High Risk Event in 5 mg Treatment Arm | Number of Subjects Experiencing a High Risk Event in Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/48 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/48 | 0/45
Other Adverse Events (participants affected / at risk) | 1/46 | 1/48 | 0/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Number of Subjects Experiencing a High Risk Event in 25 mg Treatment Arm (N=46) | Number of Subjects Experiencing a High Risk Event in 5 mg Treatment Arm (N=48) | Number of Subjects Experiencing a High Risk Event in Placebo Arm (N=45)
URI (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-05-24): https://cdn.clinicaltrials.gov/large-docs/76/NCT03462576/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/76/NCT03462576/SAP_001.pdf